CLINICAL TRIAL: NCT06876103
Title: Investigating the Effectiveness of an Online Religiously-integrated Cognitive Behavioral Therapy-based Intervention on Death Anxiety
Brief Title: Effectiveness of an Online Religiously-integrated Cognitive Behavioral Therapy-based Intervention on Death Anxiety
Acronym: RCBT-DA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Haldun University (Other)
Responsible Party: Principal Investigator, Büşra Kavla, Principal Investigator, Ibn Haldun University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/04-14
Record Dates: First submitted 2025-03-05; First posted 2025-03-14 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-03

CONDITIONS: Death Anxiety
Keywords: death anxiety; religiously integrated cognitive behavioral therapy; classical cognitive behavioral therapy; randomized control study
MeSH Terms: conditions — Necrophobia

STUDY DESIGN:
Intervention Model Description: This study employs a parallel assignment design, where participants are randomly allocated to either the intervention or control group to compare treatment effects.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to whether they are receiving religiously integrated CBT (RCBT) or classic CBT. Additionally, the outcomes assessor will be blinded to participants' pre- and post-treatment scale scores. However, the therapist conducting the intervention will be aware of the treatment allocation. Therefore, the study follows a single-blind design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Religiously Integrated CBT Group (Experimental): Participants will receive a novel online RCBT-based intervention consisting of 7 weekly 90-minute sessions in a group format.
  Interventions: Other: Religiously-integrated Cognitive Behavioral Therapy
- Classical CBT Group (Active Comparator): Participants will receive an online CBT intervention based on Furer and Walker's (2008) protocol, consisting of 7 weekly 90-minute sessions in a group format.
  Interventions: Other: Classical Cognitive Behavioral Therapy

INTERVENTIONS:
Other: Religiously-integrated Cognitive Behavioral Therapy — This study aims to assess the efficacy and feasibility of a newly developed online intervention for death anxiety based on Religiously Integrated Cognitive Behavioral Therapy (RCBT). Building upon the framework of Furer and Walker's 2008 intervention protocol, this adaptation incorporates beliefs in an afterlife, aligning with Turkish society's cultural and religious values.
  The RCBT intervention consists of seven structured group therapy sessions, each lasting 90 minutes. The program is designed to help participants identify and challenge unhelpful thoughts related to death anxiety while integrating religious resources to promote cognitive restructuring. Key components of the intervention include psychoeducation, cognitive restructuring, exposure exercises, the concept of repentance in the context of trust and belief in the afterlife, gratitude, and value-oriented behaviors.
  Arms: Religiously Integrated CBT Group
Other: Classical Cognitive Behavioral Therapy — The standard CBT intervention follows the structured protocol developed by Furer and Walker (2008), which targets cognitive distortions, avoidance behaviors, and excessive safety-seeking behaviors contributing to death anxiety. The researcher has adapted the session content to fit the protocol's core components while maintaining fidelity to the original intervention model. Sessions last 90 minutes and are conducted in an online group format.
  Session Structure: Session 1: Treatment Rationale, Session 2: Reducing Excessive Checking, Reassurance Seeking, and Safety Behaviors, Session 3: Exposure, Session 4: Cognitive Reappraisal, Session 5: Enhancing Enjoyment of Life, Session 6: Healthy Lifestyle, and Session 7: Relapse Prevention.
  Arms: Classical CBT Group

SUMMARY:
There has been growing awareness of the importance of death anxiety (DA) in pathological anxiety. DA is defined as a persistent and unreasonable fear of death and thoughts, fears, and emotions associated with the end of life. DA has been suggested as a core fear that underpins the emergence and perseverance of numerous anxiety disorders. However, previous DA-based treatment studies focus on the elderly, the patients, or health professionals who care for the terminally ill. Therefore, there is a need to examine the effect of psychological interventions on DA and current disorder symptoms in a clinical sample through randomized controlled trials. The current study aims to develop a novel Religiously Integrated Cognitive Behavioral Therapy (RCBT)-based intervention on DA in individuals diagnosed with an anxiety disorder and to compare the effectiveness of RCBT-based intervention with classical CBT-based intervention.

DETAILED DESCRIPTION:
Religion facilitates the pursuit of symbolic immortality by providing individuals with purpose and hope in both life and death. Those who believe in an afterlife also see their world as fairer, which results in lower levels of psychiatric symptoms. Previous CBT-based death anxiety interventions did not consider the assumption of an afterlife. RCBT is an approach that integrates spiritual or religious beliefs into the therapeutic process. RCBT is an approach that recognizes the importance of spirituality or religion in a client's life and aims to use these beliefs and practices positively within the context of evidence-based CBT. Briefly, no intervention studies have investigated the effect of RCBT on DA. This will be the first study to develop an RCBT-based intervention for DA.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* A score of > 26 on the Turkish Death Anxiety Scale
* Diagnosed with one of the anxiety disorders
* Believing in life after death

Exclusion Criteria:

* Diagnosed with schizophrenia, schizophreniform disorder, schizoaffective disorder, and delusional disorder
* Being in an active manic episode
* Possessing a mental disorder that interferes with completing measures or understanding the exercises conducted during sessions
* Extreme symptoms of depression (score of > 20 on the Patient Health Questionnaire (PHQ-9), and >1 on the item assessing suicidality)
* Currently receiving therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Turkish Death Anxiety Scale (TDAS) | Baseline (pretest), Week 7 (posttest), 3-month follow-up
  The Turkish Death Anxiety Scale consists of 20 items that are divided into three subscales: (a) ambiguity of death, (b) exposure to death, and (c) agony of death. These subscales exhibit strong internal consistency, with Cronbach's alpha values of .91, .94, .76 respectively, adding up to a total of .95). It consists of a five-point Likert (0 = Never to 4 = Always). Subscale scores are determined by summing the individual item scores, and the total scale score is determined by summing the subscale scores. Total scale scores can be between 0 and 80, and the higher the score, the greater the level of DA. A score range of 0-7 indicates very low-level DA, 8-25 indicates low-level DA, 26-44 indicates medium-level DA, 45-63 indicates high-level DA, and 64-80 indicates very high-level DA.
Abdel-Khalek's Death Anxiety Scale (ASDA) | Baseline (pretest), Week 7 (posttest), 3-month follow-up
  Abdel-Khalek's Death Anxiety Scale is a 20-item questionnaire that measures DA. The scale is one-dimensional. Higher scores indicate a greater degree of DA. It consists of a five-point Likert (1 = No to 5 = Very much). The Turkish reliability and validity of the scale were conducted by Sarıçiçek-Aydoğan et al. in 2015 (Cronbach's alpha = .86).

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Baseline (pretest), Week 7 (posttest), 3-month follow-up
  Generalized Anxiety Disorder-7 consists of a four-point Likert (0 = never to3 = almost every day) and 7 items that assess anxiety symptoms. The highest score that can be attained ranges up to 21. A score range of 0-4 indicates mild anxiety, 5-9 indicates moderate anxiety, 10-14 indicates high anxiety, and 15-21 indicates severe anxiety. A cut-off point of 10 points was determined for the total score. The Turkish reliability and validity of the scale were conducted by Konkan et al. in 2013 (Cronbach's alpha = .85).
Patient Health Questionnaire (PHQ-9) | Baseline (pretest), Week 7 (posttest), 3-month follow-up
  Patient Health Questionnaire consists of a four-point Likert and nine items that screen depressive symptoms. Each of these items is rated on a scale of 0 (never) to 3 (almost every day). The highest score that can be attained ranges up to 27. A score range of 1-4 indicates low depressive symptoms, 5-9 indicates mild depressive symptoms, 10-14 indicates moderate depressive symptoms, 15-19 indicates partially severe depressive symptoms, and 20-27 indicates severe depressive symptoms. The Turkish reliability and validity of the scale were conducted by Sarı et al. (2016) (Cronbach's alpha = .84).

OTHER OUTCOMES:
Belief in a Day of Judgment Scale | Baseline (pretest), Week 7 (posttest), 3-month follow-up
  The Belief in a Day of Judgment Scale comprises 20 items with two subscales: (1) belief in a day of judgment, and (2) bad behavior/actions toward others. It consists of a five-point Likert (1 = Strongly disagree to 5 = Strongly agree). Examples of the items include, "God is the savior and judge of mankind.", and "If I am pure of heart and hands, I shall live in the fear of a just God". A high score on the Belief in a Day of Judgment subscale indicates a strong belief in a Day of Judgment, the conviction that God will judge the living and the dead, and the belief in life after death. A high score on the Bad Behavior/Actions Toward Others subscale reflects the belief that human relationships and actions towards others will be scrutinized on the Day of Judgment. The Turkish reliability and validity of the scale were conducted by Turan et al. in 2020 (Cronbach's alpha = .92).
Muslim Practice and Belief Scale | Baseline (pretest), Week 7 (posttest), 3-month follow-up
  The Muslim Practice and Belief Scale- Short Form comprises nine items with two subscales: (1) social beliefs and prayers, and (2) individual beliefs and prayers subscale (PF). It consists of a five-point Likert (1 = Strongly Disagree to 5 = Strongly Agree). The Turkish reliability and validity of the scale were conducted by Akın and Yalnız in 2015 (Cronbach's alpha = .90). The subscales demonstrate good internal consistency, with Cronbach's alphas of. 86 and .91 respectively. Higher scores indicate a greater level of Muslim practice and belief.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Kavla, PhD Student, Principal Investigator — Ibn Haldun University; Burcu Uysal, Associate Professor, Study Chair — Ibn Haldun University
Locations (1):
- Ibn Haldun University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to confidentiality concerns and ethical considerations.

REFERENCES:
- [Background] Aydoğan, A. S., Gülseren, Ş., Sarıkaya, Ö. Ö., & Özen, Ç. (2015). Abdel-Khalek ölüm anksiyetesi ölçeği Türkçe formunun üniversite öğrencilerinde geçerlilik ve güvenilirliği. Nöropsikiyatri Arşivi, 52, 371-375.
- [Background] Abdel-Khalek AM. A general factor of death distress in seven clinical and non-clinical groups. Death Stud. 2004 Nov;28(9):889-98. doi: 10.1080/07481180490491040. PMID 15493083